CLINICAL TRIAL: NCT05607186
Title: Outcomes of Neoadjuvant Therapy for Rectal Cancer in a Tertiary Asian
Brief Title: Outcomes of Neoadjuvant Therapy for Rectal Cancer in a Tertiary Asian Institute
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/2342
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-10

CONDITIONS: Rectal Cancer; Oncology
MeSH Terms: conditions — Rectal Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: neoadjuvant long course chemoradiotherapy — neoadjuvant long course chemoradiotherapy consist of radiosensitizing 5FU or capecitabine and 50.4 Gy in 28 fractions over 5 weeks

SUMMARY:
This is a retrospective cohort study that aims to evaluate the correlation of magnetic resonance tumour regression grade (mrTRG) and pathological TRG (pTRG) of locally advanced rectal cancer after neoadjuvant long course chemoradiotherapy as well as the prognostic value of mrTRG on survival.

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer
* At least 1 high risk feature on MRI
* Undergo long course neoadjuvant chemoradiotherapy (LCCRT)

Exclusion Criteria:

* metastatic disease
* Patients who undergo short course radiotherapy
* Patients without a repeat MRI after completion of LCCRT

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with locally advanced rectal cancer were recruited from the Department of Colorectal Surgery, Singapore General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation between mrTRG and pTRG | Between 1 Jan 2011 to 31 Dec 2016

SECONDARY OUTCOMES:
Prognostic value of mrTRG on survival outcomes of rectal cancer patients | Between 1 Jan 2011 to 31 Dec 2016

IPD SHARING:
Plan to Share IPD: No